CLINICAL TRIAL: NCT04402047
Title: Electroacupuncture vs Topical Diclofenac Sodium Gel for Patients With Hand Osteoarthritis: Study Protocol for a Randomized Controlled Trial
Brief Title: Electroacupuncture vs Topical Diclofenac Sodium Gel for Patients With Hand Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-015-KY
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Hand Osteoarthritis
Keywords: Hand osteoarthritis; Electroacupuncture; Diclofenac sodium gel
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Efficacy evaluators and data analysts will be blinded to the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture group (Experimental)
  Interventions: Other: Electroacupuncture
- Topical DSG group (Active Comparator)
  Interventions: Drug: Topical diclofenac sodium gel

INTERVENTIONS:
Other: Electroacupuncture — We will apply Ashi points, Ex-UE9, SI3, and TE5. Sterile needles (0.3mm× 40mm) and SDZ-V EA apparatus will be utilized. Acupuncturists will insert needles perpendicularly into Ashi points for approximately 2-3mm until they pierce into the bone surface; acupuncturists will insert needles horizontally into Baxie points towards the wrist with a depth of 5-10mm; and acupuncturists will insert needles perpendicularly into SI3 and TE5 for approximately 5-10mm. All needles except Ashi points will be manually manipulated to achieve De qi. The needles at Baxie 1 and Baxie 4 will be connected using alligator clips from the EA apparatus. The electrical stimulation will last for 30 minutes with a continuous wave of 10 Hz and a fixed current intensity of 0.5 to 2 mA. All the needles will be retained for 30 minutes. Participants will undergo EA treatment three times per week for a total of 12 sessions in four consecutive weeks. If bilateral hands were affected, both sides will be treated.
  Arms: Electroacupuncture group
Drug: Topical diclofenac sodium gel — The gel will be gently rubbed over the affected joints without excessive joint movement four times per day for 4 weeks and will be asked not to wash hands for one hour after application. Each hand treatment will be used in identical dispensing doses of gel (4 cm strip, approximately 2g, which was judged sufficient for approximately half the surface of each hand (200 cm2)). Dosing times should be distributed evenly over waking hours.If bilateral hands were affected, both sides will be treated.
  Arms: Topical DSG group

SUMMARY:
Hand osteoarthritis (OA) is a prevalent joint disorder characterized by pain, stiffness, and bony enlargements/swellings of multiple joints, in particular distal interphalangeal (DIP), proximal interphalangeal (PIP) and first carpometacarpal (CMC) joints. Symptomatic hand OA is estimated to affecting 15.9% of women and 8.2% of men in the general population with a variable disease course, occurring more frequently in the elderly. Many factors including age, gender, obesity, genetic predisposition, joint deformity, joint hypermobility, and trauma are implicated in the development of hand OA. In addition to pain and stiffness, patients with hand OA often suffer from the reduced grip and pinch strength, decreased range of motion in involved and noninvolved joints, and difficulty performing dexterous tasks, resulting in disability in activities of daily living and considerable frustration.

At present, no therapies can completely cure hand OA and few therapeutic options with proven effectiveness for hand OA exist. Diclofenac sodium gel (DSG) is one of the commonly used topical NSAIDs, which can provide local pain relief for patients with hand OA with reduced systemic exposure, potentially reducing the risk of adverse events (AE). Acupuncture is effective in a host of pain-related conditions, ranging from low back pain, neck pain, shoulder pain, migraine to pain from knee OA. The research on the effects of acupuncture in people with hand OA is very limited.

The purpose of this study is to investigate the clinical effectiveness of 4-week electroacupuncture(EA) compared to topical DSG in the treatment of hand OA. Our primary hypothesis was that EA would result in a greater pain relief improvement in hand OA compared with topical DSG.

ELIGIBILITY:
Inclusion Criteria:

1. History of hand OA for at least 3 months before enrolment and use of a NASID for ≥ 1 episode of pain;
2. Reported an average possible overall finger joints pain intensity in the dominant hand over the past 48 hours of at least 40mm according to a 100-mm visual analog scale (VAS) after 1-week wash-out period of previous OA medications(Patients applying NSAIDs at the screening had to have an increase in pain in the dominant hand of ≥ 20 mm during washout);
3. Posterior-anterior radiographs had to show Kellgren-Lawrence grade 1, 2, or 3 changes in symptomatic joints;
4. Rheumatoid factor and anticyclonic citrullinated peptide were negative in all eligible participants to exclude inflammatory arthritis;
5. Ability to comply with the study protocol, understand the medical information forms as well as having signed informed consent.

Exclusion Criteria:

1. History or current evidence of secondary OA(due to causes other than a solely degenerative joint disease) or symptomatic OA at additional locations besides the hand(s) requiring treatment, or any painful syndrome of the upper limb which may interfere with evaluation of hand pain;
2. History of inflammatory arthritis(e.g., rheumatoid arthritis (RA), psoriatic arthritis), hemochromatosis, metabolic, or neuropathic arthropathies;
3. History of trauma, dislocation or operation to the hand or arm in the previous 3 months;
4. Hand pain and stiffness due to tissue scarring or tendinitis;
5. Skin damage or serious skin disorders in the hands;
6. Intake of antidepressants, anticonvulsants, vascular or narcotics during the 10 days prior to beginning the study;
7. Oral, intramuscular, intra-articular or intravenous corticosteroids, or hyaluronic acid injection within 3 months preceding enrollment;
8. Serious uncontrolled medical conditions such as cancer, uncontrolled cardiovascular disorder, severe hepatic/renal insufficiency or coagulation disorder;
9. Known allergy, contraindication or intolerance to diclofenac, acetaminophen, or gel components;
10. Known phobic to acupuncture or received acupuncture treatment within 4 weeks prior to enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in average overall finger joints pain intensity in the dominant hand over the past 48h from baseline to week 4 | at baseline and week 4
  Pain intensity will be measured using a 0-100 VAS, with 0 indicating no pain and 100 indicating maximal pain.

SECONDARY OUTCOMES:
Change in average overall finger joints pain intensity in the dominant hand over the past 48h from baseline to weeks 8, 16 | at baseline，week 8 and week 16
  Pain intensity will be measured using a 0-100 VAS, with 0 indicating no pain and 100 indicating maximal pain.
The proportion of participants achieving at least a 15-point reduction in average overall finger joints pain intensity in the dominant hand from baseline to weeks 4, 8 and 16 | at week 4, week 8 and week 16
Change in Australian Canadian Osteoarthritis Hand Index (AUSCAN) total score, and pain, stiffness and physical function subscales from baseline to weeks 4, 8 and 16 | at baseline，week 4, week 8 and week 16
  The AUSCAN index contains a 15-item scale referring to hand pain (5 items), stiffness (1 item), and function (9 items) during the preceding 48 hours, which is valid, reliable and responsive in patients with hand OA. All items are scaled on a 0-100 VAS (0=none to 100= very severe), with higher scores indicating more severe symptoms/function.
Change in Functional Index for HOA (FIHOA) from baseline to weeks 4, 8 and 16 | at baseline，week 4, week 8 and week 16
  The FIHOA is a patient-reported hand function questionnaire, comprising 10 items with a four-point Likert scale, in which 0 represents "possible without difficulty", 1 indicates "possible with slight difficulty", 2 represents "possible with important difficulty" and 3 indicates "impossible"
Change in the number of self-reported painful joints and painful joints at digital pressure from baseline to weeks 4, 8 and 16 | at baseline，week 4, week 8 and week 16
  All finger joints will be reported spontaneously for the presence of pain by the participants, and examined by a trained research nurse for the presence of pain at digital pressure.
Change in the number of swollen joints from baseline to weeks 4, 8 and 16: | at baseline，week 4, week 8 and week 16
  All soft swollen finger joints count (0-30) will be assessed by a trained research nurse at each study visit.
Change in hand grip strength and pinch strength of the fingers from baseline to weeks 4, 8 and 16: | at baseline，week 4, week 8 and week 16
  Hand grip strength and pinch strength of the fingers of the dominant hand will be tested using a hand dynamometer and a Jamar digital pinch gauge respectively.
Change in patient global assessment of improvement from baseline to weeks 4, 8 and 16 | at baseline，week 4, week 8 and week 16
  The patients will be asked to respond to the question 'Considering all the ways your hand OA affects you, how have you been during the last 48 h?' on a self-administered 0-100 VAS (0, worst possible, to 100, best possible, in 10-point increments)
The proportion of responder according to the Outcome Measures in Rheumatological Clinical Trials (OMERACT) and Osteoarthritis Research Society International (OARSI) responder criteria at weeks 4，8 and 16 | at week 4, week 8 and week 16
  The OMERACT-OARSI response is defined as an improvement in either pain (0-100 overall finger joints pain) or function (0-36 AUSCAN physical function) with ≥50% (relative) and ≥20/100 (absolute); or if the improvement is ≥20% (relative) and ≥10/100 (absolute) in ≥2 of the following: pain, functioning and patient global assessment of improvement.
Change in quality of life assessed by the World Health Organization Quality of Life abbreviated version (WHOQOL-BREF) from baseline to weeks 4, 8 and 16 | at baseline，week 4, week 8 and week 16
  The WHOQOL-BREF is a 26-item self-report questionnaire rated on a 5-point Likert-type scale with four domains of QOL: physical (seven items), psychological (six items), social (three items), and environment (eight items), plus 2 items representing the general QOL. The four domain scores are scaled in a positive direction with higher scores indicating a higher quality of life.
Self-reported consumption of acetaminophen for hand OA during weeks 1-4 and weeks 5-12 | at weeks 1-4 and weeks 5-12
  The proportion of participants using acetaminophen and the average dosage of acetaminophen used weekly will be calculated and assessed.

OTHER OUTCOMES:
Participants' expectations for acupuncture at baseline | at baseline
  At baseline, participants in the EA group will be asked to answer the following question: "What do you expect from EA treatment to improve your hand OA?"
Incidence of adverse events | weeks 1-16
  Any adverse events (AEs) during the whole study, whether reported spontaneously by the participants, or observed by the researcher, will be recorded and categorized as acupuncture-related AEs(e.g., fainting, broken needle, localized hematoma, dizziness, or), the side effect of TDG (e.g., skin irritation/itching, reddening, scaly skin), and non-treatment-related AEs. All AEs will be recorded in detail in the case report form.

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, MD, PhD, Principal Investigator — Department of Acupuncture, Guang'anmen Hospital, China Academy of Chinese Medical Sciences
Locations (1):
- Department of Acupuncture and Moxibustion, China Academy of Chinese Medical Sciences Guang'anmen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data are available on reasonable request. You can send e-mail to us if you have any question
Supporting Information: Study Protocol, SAP
Time Frame: It depends
Access Criteria: It depends

REFERENCES:
- [Derived] Wang W, Yu S, Long Z, Liu Y, Yan Y, Sun T, Liu Z. Electroacupuncture vs topical diclofenac sodium gel for patients with hand osteoarthritis: study protocol for a randomized controlled trial. J Orthop Surg Res. 2022 Apr 12;17(1):233. doi: 10.1186/s13018-022-03125-1. PMID 35413861